CLINICAL TRIAL: NCT03807661
Title: Percutaneous Deep Vein Arterialization Post-Market Study
Acronym: PROMISE UK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LimFlow SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU PMS Revision 4.4-UK
Record Dates: First submitted 2019-01-11; First posted 2019-01-17 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Critical Limb Ischemia
Keywords: Desert foot; No-option patients; Venous arterialization
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Percutaneous deep vein arterialization (Experimental): Creation of an arterio-venous fistula in the below-the-knee vasculature using the LimFlow System endovascular, minimally invasive approach
  Interventions: Procedure: Percutaneous deep vein arterialization; Device: LimFlow System

INTERVENTIONS:
Procedure: Percutaneous deep vein arterialization — Creation of an arterio-venous fistula in the below-the-knee vasculature using the LimFlow System endovascular, minimally invasive approach
Device: LimFlow System — Creation of an arterio-venous fistula in the below-the-knee vasculature using the LimFlow System endovascular, minimally invasive approach

SUMMARY:
The objective of this post-market study is to evaluate the safety and effectiveness of the LimFlow System in creating a below-the-knee arterio-venous fistula for venous arterialization in subjects with critical limb ischemia.

DETAILED DESCRIPTION:
This study will investigate the safety and effectiveness of the LimFlow System for creating an arterio-venous fistula in the below-the-knee vascular system using an endovascular, minimally invasive approach for the treatment of critical limb ischemia in subjects ineligible for conventional endovascular or surgical limb salvage procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be > 21 and < 95 years of age
* Clinical diagnosis of symptomatic critical limb ischemia, defined as Rutherford category 5 or 6
* Assessment that no conventional surgical or endovascular treatment is possible
* Proximally, the target in-flow artery at the cross-over point must be treatable with a 3.5 - 4.0 mm stent after pre-treatment (by visual estimate), and be <50% stenosed
* Subject is willing and has adequate support to comply with protocol requirements, including medication regimen and follow-up visits

Exclusion Criteria:

* Concomitant hepatic insufficiency, deep venous thrombus in target limb, uncorrected coagulation disorders, or current immunodeficiency disorder
* Prior vein stripping surgery and/or vessel harvesting for CABG in the limb intended for study
* Life expectancy less than 12 months
* Patient currently taking coumarin/warfarin which, in the opinion of the attending physician, interferes with the patient's treatment
* Any significant medical condition which, in the attending physician's opinion, may interfere with the patient's optimal treatment
* Patient currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this treatment
* Patient unable to give consent
* Pregnant or breastfeeding women
* Documented myocardial infarction or stroke within previous 90 days
* Patients suffering from renal insufficiency (GFR value less than 30 ml/min/1.73 m²) who are not on hemodialysis
* Patients with vasculitis and/or untreated popliteal aneurysms
* Patients with acute limb ischemia
* Prior peripheral arterial bypass procedure above or below the knee which could inhibit proximal inflow to the stent graft
* Lower extremity venous disease with significant edema in the target limb that may inhibit the procedure and/or jeopardize wound healing, in the investigator's opinion
* Known or suspected systemic or severe infection (e.g., WIfI foot Infection grade of 3)
* Known or suspected allergies or contraindications to stainless steel, nickel, or contrast agent that cannot be adequately pre-treated, or patients who cannot receive anticoagulation or antiplatelet aggregation therapy
* Severe heart failure, which in the opinion of the investigator may compromise subject's ability to safely undergo a percutaneous procedure (e.g., known ejection fraction of < 40%, NYHA Classification III-IV)

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - North Bristol NHS Trust, Bristol
  - Glenfield Hospital, Leicester
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 64 subjects were screened at 6 sites across England, during the time period from 11-Dec-2019 to 26-Oct-2022, yielding 28 subjects enrolled in the study.
Pre-assignment Details: Subjects were screened by site personnel and once it was deemed they met clinical inclusion and exclusion criteria, consent was obtained and angiographic and ultrasound imaging of the target arterial and venous anatomy were uploaded for review by an independent review committee. The subject was thereafter screened for suitability as an angiographically-confirmed "no option" patient who had no capacity for treatment with standard endovascular treatment or surgical bypass.
Groups:
- ITT Population: All subjects successfully screened and enrolled in the study with treatment or attempted treatment with the LimFlow System.
Period: Overall Study
Arm/Group | ITT Population
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: killograms per squared metre] | 26.1 (5.0)
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (11.2)
Current or Former Smoker [Count of Participants; unit: Participants] — Population: Smoking history unknown in 1 subject
  Participants
    number analyzed (Participants) | 27
    (all) | 21
Baseline Diabetes Status [Count of Participants; unit: Participants] | 23
Hypertension requiring medication [Count of Participants; unit: Participants] | 21
Hyperlipidaemia req. medication [Count of Participants; unit: Participants] | 16
Renal insufficiency [Count of Participants; unit: Participants]
  Any Renal Insufficiency | 5
  Renal Insufficiency Requiring Dialysis | 3
Heart Failure [Count of Participants; unit: Participants] | 7
Prior intervention to target limb [Count of Participants; unit: Participants] | 26
Rutherford classification [Count of Participants; unit: Participants] — Rutherford's chronic limb ischemia classification consists of seven (7) categories:
  * 0 Asymptomatic
  * 1 Mild claudication
  * 2 Moderate claudication
  * 3 Severe claudication
  * 4 Ischemic rest pain
  * 5 Minor tissue loss
  * 6 Major tissue loss
  Participants
    Rutherford Class 5 | 26
    Rutherford Class 6 | 2

OUTCOME MEASURES:

1. Primary Outcome: Amputation-free Survival
Description: Freedom from death or major amputation
Time Frame: Throughout one year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 28
percentage of participants | 67.2 [46.4 to 81.4]

2. Secondary Outcome: Wound Healing
Description: Complete index wound healing as assessed by wound pictures
Time Frame: Throughout one year
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 17
Participants | 12

3. Secondary Outcome: Primary and Secondary Patency
Description: Stent graft primary and secondary patency as assessed by duplex ultrasound
Time Frame: Throughout one year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 27
percentage of participants
  Primary patency | 31.7 [13.5 to 51.8]
  Secondary patency | 43.4 [22.1 to 63.1]

4. Secondary Outcome: Limb Salvage
Description: Freedom from major amputation
Time Frame: Throughout one year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 28
percentage of participants | 81.2 [60.6 to 91.8]

5. Secondary Outcome: Technical Success (Procedure Completion)
Description: Procedure completion and immediate morphological success with successful placement of the arterial and venous catheters in the desired location in the limb, and ability to place the stent graft, as assessed angiographically
Time Frame: Immediately post-procedure (approximately 4 hours after vascular access)
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 28
Participants | 27

6. Secondary Outcome: Procedural Success (Technical Success Without Death, Major Amputation, or Re-intervention)
Description: Combination of technical success without death, major amputation, or re-intervention
Time Frame: One month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Deep Vein Arterialization
Number analyzed (Participants) | 28
Participants | 20

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Percutaneous Deep Vein Arterialization
All-Cause Mortality (participants affected / at risk) | 4/28
Serious Adverse Events (participants affected / at risk) | 26/28
Other Adverse Events (participants affected / at risk) | 19/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Deep Vein Arterialization (N=28)
Arterial or venous occlusion (target limb) (Vascular disorders) | 23 (44)
Wound healing disorder (Vascular disorders) | 6 (7)
Wound infection (Infections and infestations) | 5 (5)
New wound or ulcer (Vascular disorders) | 4 (4)
Bleeding (non-target limb) (Blood and lymphatic system disorders) | 3 (3)
Gangrene or necrosis (Vascular disorders) | 3 (3)
Other blood flow abnormality (target limb) (Vascular disorders) | 3 (3)
Pain (target limb) (Vascular disorders) | 3 (3)
Chest infection (Infections and infestations) | 2 (2)
Heart failure (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2)
Sepsis or systemic infection (Infections and infestations) | 2 (2)
Access site bleeding or hematoma (Surgical and medical procedures) | 1 (1)
Anemia (Metabolism and nutrition disorders) | 1 (1)
Cardiac rhythm disorder (Cardiac disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Metabolism and nutrition disorders) | 1 (1)
Edema (Vascular disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Hypoglycemia or hyperglycemia (Endocrine disorders) | 1 (1)
Mitral valve regurgitation (Cardiac disorders) | 1 (1)
Myocardial infarction (Vascular disorders) | 1 (1)
Pain (non-target limb) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Cardiac disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Deep Vein Arterialization (N=28)
Arterial or venous occlusion (target limb) (Vascular disorders) | 6 (6)
COVID-19 (Infections and infestations) | 4 (4)
Wound infection (Infections and infestations) | 4 (4)
Bleeding (non-target limb) (Blood and lymphatic system disorders) | 3 (4)
Chest infection (Infections and infestations) | 3 (3)
Edema (Vascular disorders) | 3 (3)
Cardiac rhythm disorder (Cardiac disorders) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Hypoglycemia or hyperglycemia (Endocrine disorders) | 2 (2)
New wound or ulcer (Vascular disorders) | 2 (2)
Pain (target limb) (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
PROMISE UK was a post-market study of a CE-marked device and consisted of a single study arm with no direct comparator due to the extreme nature of the alternative other than major amputation. As such, all data reported are descriptive and are not tested in a statistical nature against the known rates of amputation and mortality of no treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT03807661/Prot_SAP_000.pdf